CLINICAL TRIAL: NCT01699087
Title: Prospective Safety and Effectiveness Study of PRK for Myopia With or Without Astigmatism Using the ALLEGRETTO WAVE® EYE-Q Excimer Laser System
Brief Title: A Safety and Effectiveness Study of PRK Using the ALLEGRETTO WAVE® EYE-Q Excimer Laser System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-10-084
Record Dates: First submitted 2012-09-27; First posted 2012-10-03 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2018-05

CONDITIONS: Myopia; Astigmatism
Keywords: PRK; myopia; astigmatism
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Photorefractive Keratectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRK ALLEGRETTO (Experimental): Photorefractive keratectomy (PRK) surgery using the ALLEGRETTO WAVE EYE-Q excimer laser system for myopic wavefront-optimized ablation
  Interventions: Procedure: Photorefractive keratectomy (PRK); Device: ALLEGRETTO WAVE EYE-Q excimer laser system

INTERVENTIONS:
Procedure: Photorefractive keratectomy (PRK) — In this corneal surgical procedure, the outer corneal epithelial layer will be removed, after which the corneal stroma will be reshaped by excimer laser ablation to reduce or eliminate refractive errors.
Device: ALLEGRETTO WAVE EYE-Q excimer laser system — The ALLEGRETTO WAVE EYE-Q excimer laser system is used for corneal stroma reshaping during PRK surgery
  Other Names: ALLEGRETTO WAVE Eye-Q; WaveLight® EX500; WaveNet™ Planning Software; ALLEGRETTO WAVE® EYE-Q excimer laser system (Model 1010-3)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the ALLEGRETTO WAVE EYE-Q excimer laser system for the reduction of myopia with or without astigmatism in subjects undergoing photorefractive keratectomy (PRK) treatment.

DETAILED DESCRIPTION:
This was a prospective, multi-center, single group study. Subjects underwent bilateral PRK in which the second eye was treated no sooner than 1 week and no later than 30 days after the first eye's PRK treatment. Subjects were followed for 2 years after surgery.

The protocol underwent 4 amendments. The key differences between the protocol versions were clarifications of the planned analyses and adverse event reporting procedures. There were no changes in the inclusion and exclusion criteria or non-adverse event related study assessments between the protocol versions 1-5.

Refractive stability of manifest refraction spherical equivalent (MRSE) and manifest refractive cylinder was defined as established when:

* At least 95% of the treated eyes had a change ≤ 1.0 diopter between manifest refractions performed at any 2 manifest refractions at least 3 months apart
* The mean rate of change, as determined by a paired analysis, was ≤ 0.5 diopter per year (0.04 D/month) over the same time period
* The mean rate of change decreased monotonically over time, with a projected asymptote of zero or a rate of change attributable to normal aging
* The 95% confidence interval for the mean rate of change included zero or a rate of change attributable to normal aging.

Refractive stability was assessed for pairs of visits within an interval and was defined to occur at the latter time point of the first interval at which stability was achieved.

In the final amendment to the protocol, 3 secondary objectives were made co-primary in response to Agency comments. All endpoints and analyses were modified to match.

ELIGIBILITY:
Inclusion Criteria:

* Subjects desiring refractive correction of myopia up to -6.00 Diopter (D) sphere with or without astigmatism 0 to -3.00 D and up to -6.00 D manifest refraction spherical equivalent (MRSE) at the spectacle plane measured by manifest refraction;
* Minimum best spectacle corrected visual acuity (BSCVA) in the treated eye of 20/25;
* Uncorrected visual acuity (UCVA) 20/40 or worse in the treated eye;
* Less than 0.75 D spherical equivalent (SE) difference between cycloplegic and manifest refractions;
* Stable refraction (within ± 0.5 D), as determined by MRSE for a minimum of 12 months prior to surgery;
* Demonstrated stable refraction for contact lens wearers, as specified in protocol;
* Signed informed consent document;
* Willing and able to comply with schedule for follow-up visits;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria

* Females who are pregnant, lactating, or planning a pregnancy during the time course of the study, or have another condition associated with the fluctuation of hormones that could lead to refractive changes;
* Participation in other clinical trials during this study;
* Acute or chronic disease or illness that would increase the operative risk or confound the outcomes of the study;
* Dry eye syndrome as determined by the short questionnaire for dry eye syndrome;
* Systemic medications that may confound the outcome of the study or increase the risk to the subject by affecting wound healing or tissue repair, including, but not limited to steroids, antimetabolites, immune response modifying drugs, etc.;
* Nystagmus or any other condition that would prevent a steady gaze during the PRK treatment or other diagnostic tests;
* Ocular condition that may predispose the subject to future complications;
* Previous intraocular or corneal surgery;
* Subjects who desire to have monovision;
* A known sensitivity to medications used for study procedures, including PRK;
* Presence or history of any condition or finding that makes the subject unsuitable as a candidate for PRK or study participation or may confound the outcome of the study, in the opinion of the Investigator;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2012-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, GCRA Surgical, Study Director — Alcon, a Novartis Company

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 8 investigative sites located in the United States.
Pre-assignment Details: Of the 176 participants enrolled, 15 did not meet inclusion and exclusion criteria and were exited prior to treatment as screen failures.
Period: Overall Study
Arm/Group | PRK ALLEGRETTO
Started | 176
Treated | 161
Completed | 152
Not Completed | 24
Not completed — Lost to Follow-up | 7
Not completed — Screen failure (prior to treatment) | 15
Not completed — Unable to make future visits | 2

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled subjects who underwent PRK surgery (intent-to-treat).
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 89
Region of Enrollment [Number; unit: participants]
  United States | 161

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes Achieving Uncorrected Visual Acuity (UCVA) of 20/40 or Better at Refractive Stability in Eyes With Best Spectacle-corrected Visual Acuity (BSCVA) of 20/20 or Better Preoperatively
Description: Visual acuity, with and without correction, was assessed monocularly using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at 4 meters under photopic conditions . The with-correction assessment was made with the manifest refraction at 4 meters.
Time Frame: Month 6 (post second eye surgery)
Population: Intent to treat (ITT)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Number analyzed (eyes) | 294
percentage of eyes | 100

2. Primary Outcome: Percentage of Eyes Achieving Manifest Refraction Spherical Equivalent (MRSE) Within ± 1.0 D of Zero at Refractive Stability
Description: Manifest refraction spherical equivalent (MRSE) is calculated as follows: sphere + 1/2 cylinder. The sphere and cylinder values are from the manifest refraction assessment. The manifest refraction assessment was conducted monocularly with the ETDRS chart at 4 meters under photopic conditions using a phoropter.
Time Frame: Month 6 (post second eye surgery)
Population: ITT
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Number analyzed (eyes) | 314
percentage of eyes | 99.7

3. Primary Outcome: Percentage of Eyes Achieving MRSE Within ± 0.5 D of Zero at Refractive Stability
Description: as for outcome 2
Time Frame: Month 6 (post second eye surgery)
Population: ITT
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Number analyzed (eyes) | 314
percentage of eyes | 93.3

4. Primary Outcome: Percentage of Eyes Achieving Manifest Refractive Cylinder Within ± 1.0 D of Zero at Refractive Stability
Description: Manifest refraction was performed monocularly under photopic lighting conditions using an ETDRS chart at 4 meters. The subject was manually refracted to his/her best correction using a phoropter.
Time Frame: Month 6 (post second eye surgery)
Population: ITT
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Number analyzed (eyes) | 314
percentage of eyes | 99.0

5. Primary Outcome: Percentage of Eyes Achieving Manifest Refractive Cylinder Within ± 0.5 D of Zero at Refractive Stability
Description: as for outcome 4
Time Frame: Month 6 (post second eye surgery)
Population: ITT
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Number analyzed (eyes) | 314
percentage of eyes | 92.7

6. Primary Outcome: Percentage of Eyes That Have a Change of ≤ 1.0 D in MRSE and Manifest Refractive Cylinder Between Consecutive Scheduled Visits
Description: MRSE is calculated as sphere + 1/2 cylinder. The sphere and cylinder values are from the manifest refraction assessment. The manifest refraction assessment was conducted monocularly with the ETDRS chart at 4 meters under photopic conditions using a phoropter.
Time Frame: Up to Month 24 (post second eye surgery)
Population: ITT
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Number analyzed (eyes) | 320
percentage of eyes
  Week 1 to Month 1 | 90.9
  Month 1 to Month 3: number analyzed (eyes) | 317
  Month 1 to Month 3 | 95.6
  Month 3 to Month 6: number analyzed (eyes) | 314
  Month 3 to Month 6 | 99.7
  Month 6 to Month 9: number analyzed (eyes) | 314
  Month 6 to Month 9 | 100
  Month 9 to Month 12: number analyzed (eyes) | 310
  Month 9 to Month 12 | 99.7
  Month 12 to Month 24: number analyzed (eyes) | 303
  Month 12 to Month 24 | 100

7. Primary Outcome: Cumulative Incidence of Ocular Serious Adverse Events by Eye
Description: Participants were followed for the duration of the study, an expected average of 24 months.
Time Frame: Up to Month 24 (post second eye surgery)
Population: ITT
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Number analyzed (eyes) | 320
eyes
  Corneal infiltrates | 2
  Corneal oedema | 1

8. Primary Outcome: Percentage of Eyes With BSCVA Decrease of ≥ 2 Lines From Baseline at Refractive Stability
Description: Visual acuity with correction was assessed monocularly using the ETDRS chart at 4 meters under photopic conditions . A decrease in 2 lines or more is considered clinically relevant (i.e. worse).
Time Frame: Month 6 (post second eye surgery)
Population: ITT
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Number analyzed (eyes) | 314
percentage of eyes | 0.0

9. Primary Outcome: Percentage of Eyes With a BSCVA Worse Than 20/40 (for Eyes With BSCVA of 20/20 or Better Preoperatively) at Refractive Stability
Description: Visual acuity with correction was assessed monocularly using the ETDRS chart at 4 meters under photopic conditions .
Time Frame: Month 6 (post second eye surgery)
Population: ITT
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Number analyzed (eyes) | 320
percentage of eyes | 0.0

10. Primary Outcome: Percentage of Eyes With > 2.0 D of Induced Manifest Refractive Cylinder Magnitude, as Compared to Baseline, at Refractive Stability
Description: Manifest refraction was performed monocularly under photopic lighting conditions using an ETDRS chart at 4 meters. The subject was manually refracted to his/her best correction using a phoropter. The cylinder value is from the manifest refraction assessment. The induced manifest refractive cylinder is the change in magnitude of cylinder compared to baseline.
Time Frame: Month 6 (post second eye surgery)
Population: ITT
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PRK ALLEGRETTO
Number analyzed (Participants) | 161
Number analyzed (eyes) | 320
percentage of eyes | 0.0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent through the duration of a subject's participation in the study (up to 29 months). AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device. AEs were obtained as solicited comments from study participants and as observations by the Investigator as outlined in the study protocol.
Groups:
- Pre-treatment: All subjects who consented to participate in the study prior to the initiation of study treatment
- PRK ALLEGRETTO: All subjects who underwent PRK surgery using the ALLEGRETTO WAVE EYE-Q excimer laser system for myopic wavefront-optimized ablation
Arm/Group | Pre-treatment | PRK ALLEGRETTO
Serious Adverse Events (participants affected / at risk) | 0/176 | 6/161
Other Adverse Events (participants affected / at risk) | 0/176 | 123/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=176) | PRK ALLEGRETTO (N=161)
Corneal infiltrates (Eye disorders) | 0 | 2
Corneal oedema (Eye disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=176) | PRK ALLEGRETTO (N=161)
Corneal opacity (Eye disorders) | 0 | 12
Diplopia (Eye disorders) | 0 | 44
Dry eye (Eye disorders) | 0 | 42
Eye pain (Eye disorders) | 0 | 63
Foreign body sensation in eyes (Eye disorders) | 0 | 82
Photophobia (Eye disorders) | 0 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study